CLINICAL TRIAL: NCT03716193
Title: Measurement of the Partial Pressure of Oxygen in Cutaneous Tumors Using Electron Paramagnetic Resonance (EPR) Oximetry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West Virginia University (Other)
Collaborators: West Virginia Clinical and Translational Science Institute (Other); Mary Babb Randolph Cancer Center at West Virginia University Hospitals (Other)
Responsible Party: Principal Investigator, Todd Tenenholz, Radiation Oncologist, Assistant Professor, West Virginia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1804069724; NCT04112342 (obsolete NCT alias)
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Skin Lesion; Skin Cancer; Skin Melanoma; Tumor Skin
MeSH Terms: conditions — Skin Neoplasms; Melanoma | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Four cohorts based on standard treatment will be given the same intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Patients who will receive definitive surgery for a primary malignancy of the skin, will have their tumor injected with India ink for tumor marking and will be given oxygen during the measurement sessions.
  Interventions: Other: Oxygen
- Cohort 2 (Experimental): Patients who will receive definitive radiation (+/- concurrent systemic therapy) for a primary malignancy of the skin, will have their tumor injected with India ink for tumor marking and will be given oxygen during the measurement sessions.
  Interventions: Other: Oxygen
- Cohort 3 (Experimental): Patients who will receive palliative radiation (+/- concurrent systemic therapy) for any tumor involving the skin, will have their tumor injected with India ink for tumor marking and will be given oxygen during the measurement sessions.
  Interventions: Other: Oxygen
- Cohort 4 (Experimental): Patients who will receive systemic therapy alone (without radiation) for any tumor involving the skin, will have their tumor injected with India ink for tumor marking and will be given oxygen during the measurement sessions.
  Interventions: Other: Oxygen

INTERVENTIONS:
Other: Oxygen — Patients will be given oxygen via a facemask during the measurement session

SUMMARY:
This protocol will take measurements of a variety of tumors involving the skin in order to assess changes in tumor oxygen from hyperoxygenation therapy and standard cancer-directed treatments, to demonstrate the clinical feasibility of using in vivo Electron Paramagnetic Resonance (EPR) Oximetry to obtain clinically useful measurements of tumor oxygen levels from cancer patients.

DETAILED DESCRIPTION:
All patients in this study will receive standard of care therapy for their cancer at the discretion of their treating physician(s). All subjects will be assigned to one of the four cohorts for which they qualify; there is no randomization and no stratification within the cohorts.

Cohort 1 - Patients who will receive definitive surgery for a primary malignancy of the skin

Cohort 2 - Patients who will receive definitive radiation (+/- concurrent systemic therapy) for a primary malignancy of the skin

Cohort 3 - Patients who will receive palliative radiation (+/- concurrent systemic therapy) for any tumor involving the skin

Cohort 4 - Patients who will receive systemic therapy alone (without radiation) for any tumor involving the skin

All patients enrolled in this study will undergo two initial measurements of their tumor oxygen level. On the first day, a small metal disc (less than 1 cm in diameter) called a SPOTChip will be placed on the surface of the tumor, and held in place using an adhesive. The patient will then be positioned (lying down or sitting) between a set of two magnets that are used to measure the oxygen level in the tumor. A small plastic oxygen detector will be placed on the skin over the tumor. These devices will be used to take a measurement of the tumor's oxygen level at baseline, then while breathing oxygen through a clear plastic facemask, and then a final time after the oxygen facemask has been removed.

After the measurements are taken, a small amount (20-50 microliters) of India ink will be injected into the tumor using a small (28-gauge) needle. The India ink will make a permanent, dark blue/black colored mark on the tumor. The ink leaves a permanent tattoo in the spot where it is injected, unless it is physically removed surgically.

The patient will return for another measurement, at least 2 days later. This measurement will use the India ink that was previously injected (described above) and there will no longer be a need to use the SPOTChip. For the India ink tumor oxygen measurement a small piece of wire (called a loop resonator) will be placed over the tumor and held in place using medical honey and saran wrap or tape. The Investigator will first take a measurement of the tumor's oxygen level at baseline, then while breathing oxygen through a clear plastic facemask, and then the mask will be taken the tumor's oxygen level will be measured as it returns to baseline.

Patients who have surgical excision of the tumor (cohort 1) will not have any further measurements after this point.

Patients who are being treated with radiation therapy (cohorts 2 & 3), will come back for weekly measurements of the tumor during treatment, followed by one additional measurement one month after they have completed the course of radiation therapy.

Patients being treated with chemotherapy, immunotherapy, or other systemic therapies without radiation (cohort 4), will come back for measurements every 3-4 weeks around the time of their regular infusion, followed by one additional measurement one month after they complete the course of systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathology-proven (histology or cytology) malignancy of any histology and site of origin
* Visible tumor (primary or metastasis) involving the skin of at least 6 mm in diameter
* Negative serum or urine pregnancy test within 72 hours prior to registration for women of childbearing potential

Exclusion Criteria:

* Implanted electric, magnetic or mechanically activated devices like a pacemaker, defibrillator, nerve stimulator, cochlear implant or portable infusion pump. Also individuals who have any non-MRI compatible implants
* Individuals who have a ferromagnetic foreign body located in their body
* Prior adverse reaction to a charcoal product (e.g., a local hypersensitive response from a black tattoo or from ingestion of activated charcoal)
* Prior adverse reaction to gum Arabic, which is an ingredient in the India ink
* Prior allergic reaction to medical adhesives
* Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women. There is no known harm to the woman or her fetus from participating; this is precautionary only

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Assess the change in oxygenation of cutaneous tumors from hyperoxygenation therapy during the standard therapy for the disease | From the first oxygen measurement to one month after the completing standard therapy
  Tumor oxygen kinetics will be measured by EPR oximetry under ambient conditions, during hyperoxygenation therapy (100% O2 administered via a non-rebreather face mask), and immediately after hyperoxygenation therapy.

SECONDARY OUTCOMES:
To characterize temporal variations in oxygenation of cutaneous tumors over a course of local radiation therapy and/or systemic chemotherapy or immunotherapy | From the first oxygen measurement to one month after the completing standard therapy
  Patients will undergo weekly tumor oxygen measurements by EPR during a radiation therapy course and every 3-4 week measurements during cycles of systemic therapy. Changes in tumor oxygen will be correlated with standard measures of response to therapy using RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Tenenholz, MD, Principal Investigator — West Virginia University
Locations (1):
- Todd Tenenholz, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT03716193/ICF_000.pdf